CLINICAL TRIAL: NCT00996307
Title: Pivotal, Multicenter, Observer-Blind, Randomized Study of Influenza A (H1N1) 2009 Monovalent Subunit Vaccine With and Without Adjuvant in Children Ages 6 to <36 Months
Brief Title: Pivotal, Multicenter, Observer-Blind, Randomized Study of Influenza A (H1N1)2009 Monovalent Subunit Vaccine With and Without Adjuvant in Children Ages 6 to <36 Months
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V112_06
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Results first posted 2011-05-25 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Influenza
Keywords: Swine Flu; Flu; Vaccine; Children; Adjuvant; A/H1N1 2009 Influenza
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 3.75_(50)MF59 (Experimental): 3.75 µg A/H1N1 antigen with 50% MF59 adjuvant administered on study day 1 and day 22.
  Interventions: Biological: MF59-eH1N1_f
- 7.5_(0)MF59 (Experimental): 7.5 µg A/H1N1 antigen without MF59 adjuvant administered on study day 1 and day 22.
  Interventions: Biological: MF59-eH1N1_f
- 7.5_(50)MF59 (Experimental): 7.5 µg A/H1N1 antigen with 50% MF59 adjuvant administered on study day 1 and day 22.
  Interventions: Biological: MF59-eH1N1_f
- 15_(0)MF59 (Experimental): 15 µg A/H1N1 antigen without MF59 adjuvant administered on study day 1 and day 22.
  Interventions: Biological: MF59-eH1N1_f

INTERVENTIONS:
Biological: MF59-eH1N1_f — 3.75 µg A/H1N1 antigen with 50% MF59 adjuvant administered on study day 1 and day 22.
  Arms: 3.75_(50)MF59
Biological: MF59-eH1N1_f — 7.5 µg A/H1N1 antigen without MF59 adjuvant administered on study day 1 and day 22.
  Arms: 7.5_(0)MF59
Biological: MF59-eH1N1_f — 15 µg A/H1N1 antigen without MF59 adjuvant administered on study day 1 and day 22.
  Arms: 15_(0)MF59
Biological: MF59-eH1N1_f — 7.5 µg A/H1N1 antigen with 50% MF59 adjuvant administered on study day 1 and day 22.
  Arms: 7.5_(50)MF59

SUMMARY:
This study will evaluate the safety and immunogenicity of different combinations of A/H1N1 2009 (swine flu) vaccine in healthy young children

ELIGIBILITY:
Inclusion Criteria:

* Children 6 to 35 months of age in good health as determined by medical history, physical assessment and clinical judgement of the investigator and without influenza within the past 6 months

Exclusion Criteria:

* History of serious disease.
* History of serious reaction following administration of vaccine or hypersensitivity to vaccine components.
* Known or suspected impairment/alteration of immune function.
* Receipt or planned receipt of seasonal trivalent influenza vaccine within 1 week before or after each study vaccination

For additional entry criteria, please refer to protocol

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 654 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Director — Novartis
Locations (29):
- United States (28):
  - Bentonville, Arkansas
  - Fort Smith, Arkansas
  - Canoga Park, California
  - Dinuba, California
  - Fresno, California
  - Long Beach, California
  - Los Angeles, California
  - Madera, California
  - Torrance, California
  - New Albany, Indiana
  - Newton, Kansas
  - Wichita, Kansas
  - Bardstown, Kentucky
  - Woburn, Massachusetts
  - Fargo, North Dakota
  - Dayton, Ohio
  - Huber Heights, Ohio
  - Oklahoma City, Oklahoma
  - Charleston, South Carolina
  - Spartanburg, South Carolina
  - Lebanon, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Provo, Utah
  - South Jordan, Utah
  - St. George, Utah
  - West Jordan, Utah
  - Charlottesville, Virginia
- Tlalpan, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 29 sites in USA and Mexico. Five subjects received wrong vaccination according to the randomization and were excluded from PPS but were included in the safety set.
Pre-assignment Details: All subjects enrolled were included in the trial. The data entered is for the overall study.
Period: Overall Study
Arm/Group | 3.75_(50)MF59 | 7.5_(0)MF59 | 7.5_(50)MF59 | 15_(0)MF59
Started | 164 | 165 | 160 | 165
Completed | 144 | 148 | 146 | 144
Not Completed | 20 | 17 | 14 | 21
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 5 | 5
Not completed — Lost to Follow-up | 13 | 13 | 7 | 15
Not completed — Administrative reason | 0 | 1 | 0 | 0
Not completed — Unable to classify | 4 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3.75_(50)MF59 | 7.5_(0)MF59 | 7.5_(50)MF59 | 15_(0)MF59 | Total
Number analyzed (Participants) | 164 | 165 | 160 | 165 | 654
Age, Continuous [Mean (Standard Deviation); unit: Months]
  6 to <36 Months age | 21.2 (7.9) | 21.6 (8.8) | 21.1 (8.4) | 21.3 (8.9) | 21.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 79 | 80 | 78 | 312
  Male | 89 | 86 | 80 | 87 | 342

OUTCOME MEASURES:

1. Primary Outcome: Antibody Responses After the First and Second Vaccinations
Description: CBER guidance (<65 years of age): The lower bound of the two-sided 95% CI for the percent of subjects achieving seroconversion for HI antibody should be ≥ 40% AND the lower bound of the two sided 95% CI for the percent of subjects achieving an HI antibody titer ≥ 1:40 should be ≥ 70%.
Time Frame: 21 days after each vaccination
Population: The analysis was done on the per-protocol set (PPS).
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 3.75_(50)MF59 | 7.5_(0)MF59 | 7.5_(50)MF59 | 15_(0)MF59
Number analyzed (Participants) | 129 | 124 | 126 | 129
Percentages of Subjects
  HI titer ≥1:40 (Baseline) | 19 [12 to 26] | 9 [5 to 15] | 15 [9 to 23] | 19 [13 to 27]
  HI titer ≥1:40 (Day 22) | 79 [71 to 86] | 37 [29 to 46] | 86 [78 to 91] | 50 [41 to 59]
  Seroconversion Day 22 | 74 [65 to 81] | 32 [24 to 41] | 80 [72 to 87] | 44 [35 to 53]
  HI titer ≥1:40 (Day 43) | 100 [97 to 100] | 70 [61 to 78] | 100 [97 to 100] | 81 [74 to 88]
  Seroconversion Day 43 | 98 [93 to 100] | 68 [59 to 76] | 98 [94 to 100] | 76 [68 to 83]
  HI titer ≥1:40 (Day 202;N=45,38,46,38) | 96 [85 to 99] | 50 [33 to 67] | 100 [92 to 100] | 55 [38 to 71]
  Seroconversion Day 202;N=45,38,46,38) | 89 [76 to 96] | 50 [33 to 67] | 91 [79 to 98] | 39 [24 to 57]
  HI titer ≥1:40 (Day 387;N=46,37,38,36) | 85 [71 to 94] | 27 [14 to 44] | 84 [69 to 94] | 36 [21 to 54]
  Seroconversion Day 387;N=45,38,46,38) | 76 [61 to 87] | 22 [10 to 38] | 76 [60 to 89] | 25 [12 to 42]

2. Secondary Outcome: Immunogenicity Measurement by Geometric Mean Titers (GMT)
Description: Immunogenicity was measured in terms of the GMT at 21 days after each vaccination.
Time Frame: 21 days after each vaccination
Population: The analysis was done on the Full Analysis Set (FAS).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3.75_(50)MF59 | 7.5_(0)MF59 | 7.5_(50)MF59 | 15_(0)MF59
Number analyzed (Participants) | 129 | 124 | 126 | 129
Titers
  GMT Baseline | 10 [7.94 to 14] | 7.27 [5.5 to 9.6] | 9.29 [7.06 to 12] | 11 [8.22 to 14]
  GMT Day 22 | 83 [56 to 123] | 20 [14 to 31] | 92 [62 to 136] | 37 [25 to 55]
  GMT Day 43 | 642 [468 to 879] | 80 [58 to 110] | 626 [457 to 858] | 151 [110 to 206]
Statistical Analysis 1: Comparison: 3.75_(50)MF59 vs 7.5_(0)MF59; Test type: Non-Inferiority or Equivalence — The two-sided confidence intervals (CIs) were calculated and assessed for non-inferiority first against the margin of 0.5 (exploratory margin) and in case of success against the margin of 0.667 (based on CBER guidance against the licensed comparator); Ratio of GMTs = 4.06, 95% CI 2-sided [2.55 to 6.46] — Ratio of GMTs at Day 22
Statistical Analysis 2: Comparison: 3.75_(50)MF59 vs 15_(0)MF59; Test type: Non-Inferiority or Equivalence — The two-sided CIs were calculated and assessed for non-inferiority first against the margin of 0.5 (exploratory margin) and in case of success against the margin of 0.667 (based on CBER guidance against the licensed comparator); Ratio of GMTs = 2.25, 95% CI 2-sided [1.42 to 3.56] — Ratio of GMTs at Day 22
Statistical Analysis 3: Comparison: 7.5_(0)MF59 vs 7.5_(50)MF59; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; Ratio of GMTs = 4.49, 95% CI 2-sided [2.8 to 7.19] — Ratio of GMTs at Day 22
Statistical Analysis 4: Comparison: 7.5_(50)MF59 vs 15_(0)MF59; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; Ratio of GMTs = 2.49, 95% CI 2-sided [1.56 to 3.96] — Ratio of GMTs at Day 22
Statistical Analysis 5: Comparison: 3.75_(50)MF59 vs 7.5_(0)MF59; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; Ratio of GMTs = 8.01, 95% CI 2-sided [5.52 to 12] — Ratio of GMTs at Day 43
Statistical Analysis 6: Comparison: 3.75_(50)MF59 vs 15_(0)MF59; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; Ratio of GMTs = 4.25, 95% CI 2-sided [2.94 to 6.15] — Ratio of GMTs at Day 43
Statistical Analysis 7: Comparison: 7.5_(0)MF59 vs 7.5_(50)MF59; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; Ratio of GMTs = 7.81, 95% CI 2-sided [5.36 to 11] — Ratio of GMTs at Day 43
Statistical Analysis 8: Comparison: 7.5_(50)MF59 vs 15_(0)MF59; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; Ratios of GMTs = 4.15, 95% CI 2-sided [2.86 to 6.02] — Ratio of GMTs at Day 43
Statistical Analysis 9: Comparison: 3.75_(50)MF59 vs 7.5_(0)MF59; Superiority of the adjuvanted vaccines against the non-adjuvanted vaccines was to be tested against the margin of 1 on day 22; Test type: Superiority or Other; Ratio of GMTs = 3.66, 95% CI 2-sided [2.37 to 5.65]
Statistical Analysis 10: Comparison: 3.75_(50)MF59 vs 15_(0)MF59; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; Ratio of GMTs = 2.21, 95% CI 2-sided [1.43 to 3.4]
Statistical Analysis 11: Comparison: 7.5_(0)MF59 vs 7.5_(50)MF59; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; Ratio of GMTs = 4.42, 95% CI 2-sided [2.85 to 6.86]
Statistical Analysis 12: Comparison: 7.5_(50)MF59 vs 15_(0)MF59; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; Ratio of GMTs = 2.67, 95% CI 2-sided [1.72 to 4.13]
Statistical Analysis 13: Comparison: 3.75_(50)MF59 vs 7.5_(0)MF59; Superiority of the adjuvanted vaccines against the non-adjuvanted vaccines was to be tested against the margin of 1 on day 43; Test type: Superiority or Other; Ratio of GMTs = 7.82, 95% CI 2-sided [5.54 to 11]
Statistical Analysis 14: Comparison: 3.75_(50)MF59 vs 15_(0)MF59; Superiority of the adjuvanted vaccines against the non-adjuvanted vaccines; Test type: Superiority or Other; Ratio of GMTs = 4.55, 95% CI 2-sided [3.23 to 6.42]
Statistical Analysis 15: Comparison: 7.5_(0)MF59 vs 7.5_(50)MF59; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; Ratio of GMTs = 7.52, 95% CI 2-sided [5.3 to 11]
Statistical Analysis 16: Comparison: 7.5_(50)MF59 vs 15_(0)MF59; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; Ratio of GMTs = 4.37, 95% CI 2-sided [3.09 to 6.19]

3. Primary Outcome: Number of Participants Reporting Solicited Local and Systemic Reactions After First Vaccination
Description: Safety was measured in terms of the number of participants reporting solicited local and systemic reactions after first vaccination.
Time Frame: Day 1 to 7
Population: The analysis was done on the safety set which included the five subjects who received wrong vaccination according to the randomization. These five subjects were excluded from PPS.
Measure: Number; unit: Participants
Arm/Group | 3.75_(50)MF59 | 7.5_(0)MF59 | 7.5_(50)MF59 | 15_(0)MF59
Number analyzed (Participants) | 161 | 161 | 161 | 163
Participants
  Ecchymosis | 0 | 0 | 0 | 0
  Erythema | 1 | 0 | 2 | 1
  Swelling | 6 | 9 | 4 | 6
  Induration | 8 | 8 | 13 | 8
  Tenderness | 49 | 42 | 53 | 42
  Sleepiness | 36 | 28 | 38 | 30
  Diarrhea | 32 | 28 | 37 | 25
  Vomiting | 13 | 10 | 12 | 10
  Irritability | 40 | 39 | 45 | 41
  Change in eating habits | 21 | 16 | 19 | 18
  Persist crying | 34 | 35 | 35 | 35
  Fever≥38.5°C | 5 | 5 | 9 | 7

4. Primary Outcome: Number of Participants Reporting Solicited Local and Systemic Reactions After Second Vaccination
Description: Safety was measured in terms of the number of participants reporting solicited local and systemic reactions after second vaccination.
Time Frame: Day 22 to 28
Population: The analysis was done on the safety set. Almost all the subjects across the vaccine groups received their first and second vaccinations within the protocol-specified window. While all the enrolled subjects received their first vaccination, 3% to 7% of subjects across the vaccine groups did not receive their second vaccination.
Measure: Number; unit: Participants
Arm/Group | 3.75_(50)MF59 | 7.5_(0)MF59 | 7.5_(50)MF59 | 15_(0)MF59
Number analyzed (Participants) | 155 | 148 | 157 | 157
Participants
  Ecchymosis | 0 | 0 | 1 | 0
  Erythema | 1 | 1 | 4 | 1
  Swelling | 2 | 1 | 8 | 6
  Induration | 4 | 3 | 12 | 9
  Tenderness | 35 | 27 | 37 | 32
  Sleepiness | 28 | 21 | 20 | 17
  Diarrhea | 20 | 19 | 20 | 15
  Vomiting | 11 | 9 | 14 | 5
  Irritability | 36 | 39 | 32 | 24
  Change in eating habits | 20 | 18 | 14 | 11
  Persist crying | 21 | 22 | 24 | 18
  Fever≥38.5°C | 8 | 5 | 4 | 7

5. Secondary Outcome: Antibody Responses With and Without Seasonal Influenza Vaccination for Year 2009 to 2010
Description: Subgroup analysis based on receipt of recent seasonal vaccination. Comparison between subjects previously vaccinated versus not vaccinated with seasonal influenza vaccines.
Time Frame: Day 22 (three weeks after first vaccination); day 43 (three weeks after second vaccination)
Population: The analysis was done on the subgroup of the per-protocol set(PPS).
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Groups:
- 3.75_(50)MF59- No Previous Vaccination; 3.75_(50)MF59-Previous Vaccination: 3.75 µg A/H1N1 antigen with 50% MF59 adjuvant administered on study day 1 and day 22.
- 7.5_(0)MF59 - No Previous Vaccination; 7.5_(0)MF59-Previous Vaccination: 7.5 µg A/H1N1 antigen without MF59 adjuvant administered on study day 1 and day 22.
- 7.5_(50)MF59-No Previous Vaccination; 7.5_(50) MF59-Previous Vaccinaiton: 7.5 µg A/H1N1 antigen with 50% MF59 adjuvant administered on study day 1 and day 22.
- 15_(0)MF59 - No Previous Vaccination; 15_(0)MF59-Previous Vaccination: 15 µg A/H1N1 antigen without MF59 adjuvant administered on study day 1 and day 22.
Arm/Group | 3.75_(50)MF59- No Previous Vaccination | 7.5_(0)MF59 - No Previous Vaccination | 7.5_(50)MF59-No Previous Vaccination | 15_(0)MF59 - No Previous Vaccination | 3.75_(50)MF59-Previous Vaccination | 7.5_(0)MF59-Previous Vaccination | 7.5_(50) MF59-Previous Vaccinaiton | 15_(0)MF59-Previous Vaccination
Number analyzed (Participants) | 81 | 83 | 92 | 89 | 48 | 41 | 34 | 40
Percentages of Subjects
  Seroconversion (Day 22/Day 1) | 73 [62 to 82] | 37 [27 to 49] | 78 [68 to 86] | 44 [33 to 55] | 75 [60 to 86] | 22 [11 to 38] | 85 [69 to 95] | 45 [29 to 62]
  Seroconversion (Day 43/Day 1) | 99 [93 to 100] | 66 [55 to 76] | 98 [92 to 100] | 78 [67 to 86] | 96 [86 to 99] | 71 [54 to 84] | 100 [90 to 100] | 73 [56 to 85]
  HI titer ≥1:40 (Day 1) | 25 [16 to 36] | 12 [6 to 21] | 16 [9 to 25] | 21 [13 to 31] | 8 [2 to 20] | 2 [0.062 to 13] | 12 [3 to 27] | 15 [6 to 30]
  HI titer ≥1:40 (Day 22) | 78 [67 to 86] | 42 [31 to 54] | 84 [75 to 91] | 49 [39 to 60] | 81 [67 to 91] | 27 [14 to 43] | 91 [76 to 98] | 50 [34 to 66]
  HI titer ≥1:40 (Day 43) | 100 [96 to 100] | 67 [56 to 77] | 100 [96 to 100] | 83 [74 to 90] | 100 [93 to 100] | 76 [60 to 88] | 100 [90 to 100] | 78 [62 to 89]

6. Secondary Outcome: Geometric Mean Titers (GMTs) With and Without Seasonal Influenza Vaccination for Year 2009 to 2010
Description: as for outcome 5
Time Frame: Day 22 (three weeks after first vaccination); day 43 (three weeks after second vaccination)
Population: The analysis was done on the subgroup on the per-protocol set (PPS).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- 7.5_(50)MF59 - No Previous Vaccination; 7.5_(50) MF59-Previous Vaccinaiton: 7.5 µg A/H1N1 antigen with 50% MF59 adjuvant administered on study day 1 and day 22.
- 15_(0)MF59-with Previous Vaccination: 15 µg A/H1N1 antigen without MF59 adjuvant administered on study day 1 and day 22.
Arm/Group | 3.75_(50)MF59- No Previous Vaccination | 7.5_(0)MF59 - No Previous Vaccination | 7.5_(50)MF59 - No Previous Vaccination | 15_(0)MF59 - No Previous Vaccination | 3.75_(50)MF59-Previous Vaccination | 7.5_(0)MF59-Previous Vaccination | 7.5_(50) MF59-Previous Vaccinaiton | 15_(0)MF59-with Previous Vaccination
Number analyzed (Participants) | 81 | 83 | 92 | 89 | 48 | 41 | 34 | 40
Titers
  Day 1 | 11 [7.66 to 16] | 7.95 [5.58 to 11] | 9.94 [6.93 to 14] | 12 [8.3 to 17] | 10 [6.84 to 15] | 6.52 [4.28 to 9.94] | 8.30 [5.75 to 13] | 10 [6.58 to 15]
  Day 22 | 101 [61 to 167] | 25 [15 to 41] | 105 [63 to 173] | 42 [26 to 68] | 80 [43 to 148] | 17 [8.88 to 34] | 100 [51 to 194] | 45 [23 to 87]
  Day 43 | 975 [663 to 1432] | 103 [71 to 149] | 788 [538 to 1154] | 186 [129 to 271] | 389 [226 to 669] | 57 [32 to 103] | 483 [269 to 867] | 124 [69 to 224]

7. Secondary Outcome: Antibody Response Based on Baseline Seropositivity
Description: Subgroup analysis based on Subjects with a pre-vaccination HI antibody titer < 1:10 and prevaccination HI antibody titer ≥ 1:10
Time Frame: Day 22 (three weeks after first vaccination); day 43 (three weeks after second vaccination)
Population: The analysis was done on the subgroup of the per-protocol set (PPS).
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Groups:
- 3.75_(50)MF59- Baseline HI <1:10; 3.75_(50)MF59 - Baseline HI ≥1:10: 3.75 µg A/H1N1 antigen with 50% MF59 adjuvant administered on study day 1 and day 22.
- 7.5_(0)MF59 - HI <1:10; 7.5_(0)MF59 - Baseline HI ≥1:10: 7.5 µg A/H1N1 antigen without MF59 adjuvant administered on study day 1 and day 22.
- 7.5_(50)MF59 - HI <1:10; 7.5_(50)MF59 - Baseline HI ≥1:10: 7.5 µg A/H1N1 antigen with 50% MF59 adjuvant administered on study day 1 and day 22.
- 15_(0)MF59 - HI <1:10; 15_(0)MF59 - Baseline HI ≥1:10: 15 µg A/H1N1 antigen without MF59 adjuvant administered on study day 1 and day 22.
Arm/Group | 3.75_(50)MF59- Baseline HI <1:10 | 7.5_(0)MF59 - HI <1:10 | 7.5_(50)MF59 - HI <1:10 | 15_(0)MF59 - HI <1:10 | 3.75_(50)MF59 - Baseline HI ≥1:10 | 7.5_(0)MF59 - Baseline HI ≥1:10 | 7.5_(50)MF59 - Baseline HI ≥1:10 | 15_(0)MF59 - Baseline HI ≥1:10
Number analyzed (Participants) | 90 | 96 | 91 | 90 | 39 | 28 | 35 | 39
Percentages of Subjects
  Seroconversion (Day 22/Day 1) | 72 [62 to 81] | 31 [22 to 42] | 82 [73 to 90] | 39 [29 to 50] | 77 [61 to 89] | 36 [19 to 56] | 74 [57 to 88] | 56 [40 to 72]
  Seroconversion (Day 43/Day 1) | 100 [96 to 100] | 67 [56 to 76] | 100 [96 to 100] | 77 [67 to 85] | 92 [79 to 98] | 71 [51 to 87] | 94 [81 to 99] | 74 [58 to 87]
  HI titer ≥1:40 (Day 1) | 0 [0 to 4] | 0 [0 to 4] | 0 [0 to 4] | 0 [0 to 4] | 62 [45 to 77] | 39 [22 to 59] | 54 [37 to 71] | 64 [47 to 79]
  HI titer ≥1:40 (Day 22) | 72 [62 to 81] | 31 [22 to 42] | 82 [73 to 90] | 39 [29 to 50] | 95 [83 to 99] | 57 [37 to 76] | 94 [81 to 99] | 74 [58 to 87]
  HI titer ≥1:40 (Day 43) | 100 [96 to 100] | 67 [56 to 76] | 100 [96 to 100] | 77 [67 to 85] | 100 [91 to 100] | 82 [63 to 94] | 100 [90 to 100] | 92 [79 to 98]

8. Secondary Outcome: Geometric Mean Titers (GMTs) Based on Baseline Seropositivity
Description: Subgroup analysis based on Subjects with a pre-vaccination HI antibody titer < 1:10 and prevaccination HI antibody titer ≥ 1:10 Immunogenicity responses in subjects who are seropositive (A/H1N1 2009 HI titer ≥ 1:10) at Baseline (Day 1 (pre-vaccination)) as compared to those who are seronegative (HI titer < 1:10).
Time Frame: Day 22 (three weeks after first vaccination); day 43 (three weeks after second vaccination)
Population: The analysis was done on the subgroup of the per-protocol set (PPS).
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | 3.75_(50)MF59- Baseline HI <1:10 | 7.5_(0)MF59 - HI <1:10 | 7.5_(50)MF59 - HI <1:10 | 15_(0)MF59 - HI <1:10 | 3.75_(50)MF59 - Baseline HI ≥1:10 | 7.5_(0)MF59 - Baseline HI ≥1:10 | 7.5_(50)MF59 - Baseline HI ≥1:10 | 15_(0)MF59 - Baseline HI ≥1:10
Number analyzed (Participants) | 90 | 96 | 91 | 90 | 39 | 28 | 35 | 39
Titres
  Day 1 | 5.06 [4.98 to 5.14] | 5.07 [4.99 to 5.15] | 5.01 [4.93 to 5.09] | 5.06 [4.98 to 5.14] | 53 [34 to 83] | 35 [21 to 58] | 47 [29 to 76] | 69 [44 to 108]
  Day 22 | 42 [29 to 61] | 15 [11 to 22] | 60 [42 to 88] | 17 [12 to 24] | 266 [137 to 517] | 67 [31 to 145] | 313 [154 to 639] | 248 [126 to 487]
  Day 43 | 566 [398 to 804] | 65 [46 to 93] | 577 [404 to 825] | 96 [67 to 137] | 660 [390 to 1117] | 167 [90 to 308] | 811 [462 to 1426] | 420 [246 to 717]

9. Secondary Outcome: Antibody Persistence by Geometric Mean Titers (GMT)
Description: Immunogenicity was assessed in terms of Geometric Mean Titers (GMT at 6 months (Day 202)and 12 months (Day 387) after second vaccination.
Time Frame: 6 months (Day 202) and 12 months (Day 387) after second vaccination
Population: The analysis was done on the subgroup of the per-protocol set (PPS).
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 3.75_(50)MF59 | 7.5_(0)MF59 | 7.5_(50)MF59 | 15_(0)MF59
Number analyzed (Participants) | 129 | 124 | 126 | 129
Titer
  GMT (Day 1) | 10 [7.94 to 14] | 7.27 [5.5 to 9.6] | 9.29 [7.06 to 12] | 11 [8.2 to 14]
  GMT (Day 202, N=45, 38, 46, 38) | 176 [111 to 280] | 33 [20 to 54] | 205 [133 to 316] | 42 [25 to 69]
  GMT (Day 387, N= 46, 37, 38, 36) | 92 [52 to 162] | 15 [8.24 to 28] | 85 [48 to 151] | 25 [13 to 46]

ADVERSE EVENTS:
Time Frame: Throughout the entire study period. Five subjects received wrong vaccination according to the randomization and were excluded from PPS but were included in the safety set.
Description: Local, systemic, and other reactions were collected from Study days 1 to 7 and 22 to 28. SAEs, medically attended visits, new onset of chronic diseases and AEs that lead to subject's withdrawal were collected from Day 1 (post-consent) through Day 387 (12 months following second vaccination).
Arm/Group | 3.75_(50)MF59 | 7.5_(0)MF59 | 7.5_(50)MF59 | 15_(0)MF59
Serious Adverse Events (participants affected / at risk) | 5/162 | 6/164 | 1/162 | 10/166
Other Adverse Events (participants affected / at risk) | 144/162 | 152/164 | 141/162 | 142/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3.75_(50)MF59 (N=162) | 7.5_(0)MF59 (N=164) | 7.5_(50)MF59 (N=162) | 15_(0)MF59 (N=166)
Intussusception (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Abdominal abcess (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 1 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Accidental exposure to product (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Complex partial seizures (Nervous system disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Genital abscess (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3.75_(50)MF59 (N=162) | 7.5_(0)MF59 (N=164) | 7.5_(50)MF59 (N=162) | 15_(0)MF59 (N=166)
Ear pain (Ear and labyrinth disorders) | 9 | 4 | 7 | 5
Conjunctivitis (Infections and infestations) | 27 | 22 | 18 | 22
Diarrhoea (Gastrointestinal disorders) | 57 | 52 | 63 | 45
vomiting (Gastrointestinal disorders) | 33 | 37 | 33 | 24
Irritability (Psychiatric disorders) | 58 | 62 | 60 | 52
Pyrexia (General disorders) | 53 | 52 | 54 | 53
Bronchiolitis (Infections and infestations) | 10 | 12 | 9 | 13
Bronchitis (Infections and infestations) | 5 | 6 | 9 | 7
Croup infections (Infections and infestations) | 11 | 12 | 7 | 12
Ear infection (Infections and infestations) | 5 | 10 | 6 | 8
Gastroenteritis (Infections and infestations) | 12 | 9 | 4 | 8
Nasopharyngitis (Infections and infestations) | 23 | 20 | 13 | 20
Otitis media (Infections and infestations) | 56 | 38 | 37 | 45
Otitis media acute (Infections and infestations) | 14 | 10 | 12 | 12
Pharyngitis (Infections and infestations) | 18 | 16 | 12 | 17
Pharyngitis streptococcal (Infections and infestations) | 7 | 7 | 10 | 5
Rhinitis (Infections and infestations) | 14 | 11 | 13 | 13
Sinusitis (Infections and infestations) | 11 | 16 | 8 | 13
Upper respiratory tract infection (Infections and infestations) | 62 | 54 | 51 | 64
Viral infection (Infections and infestations) | 18 | 14 | 12 | 17
Crying (General disorders) | 47 | 46 | 48 | 42
Somnolence (Nervous system disorders) | 51 | 41 | 48 | 39
Eating disorder (Psychiatric disorders) | 33 | 30 | 30 | 23
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 10 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 45 | 54 | 46 | 54
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 11 | 14 | 11
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 8 | 10 | 5 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 26 | 24 | 27 | 32
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 10 | 12 | 8 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 5 | 9
Injection site pain (Nervous system disorders) | 60 | 51 | 60 | 50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No